CLINICAL TRIAL: NCT05214560
Title: Prospective Clinical Evaluation of BD Spinal Needles
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Other Study IDs: MDS-20EPSPEU001
Record Dates: First submitted 2022-01-12; First posted 2022-01-28 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Analgesia; Anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Participants who require a BD Spinal needle
  Interventions: Device: Spinal needle

INTERVENTIONS:
Device: Spinal needle — Insertion of a spinal needle to perform the neuraxial procedure.

SUMMARY:
Post-market, observational study to assess the real-world safety and efficacy of BD Spinal Needles used in an on-market fashion.

DETAILED DESCRIPTION:
Single-arm, post-market, observational, prospective study of participants who will receive neuraxial procedures with a BD Spinal Needle as part of their routine medical care.

Patients will be followed from BD Spinal needle insertion up to 7 days after the insertion according to the routine medical care and site policy.

Data collected will be gathered from the patient's medical charts.

ELIGIBILITY:
Inclusion Criteria:

* Any patient, regardless of age or gender, for which the investigator has decided that a neuraxial procedure must be performed utilizing BD Spinal Needles as part of their routine medical care
* Expected to be available for observation through the study period (7-days post procedure)
* Provision of signed and dated informed consent form (Note: Consent of guardian or parent may be required for patients under the age of 18 years; participant assent may be required as well.)

Exclusion Criteria:

* Undergoing emergency surgery
* Coagulopathy or bleeding disorder for which regional anesthesia poses an increased risk
* History of neurological impairment or disease of the trunk or lower extremities.
* Infection at or near the site of needle insertion
* Previous spine surgery at the level involved in the study procedure

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any participants who require a spinal needle device as part of their routine medical care.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Hoerauf, MD, Study Director — Becton, Dickinson and Company
Locations (6):
- Medizinische Universität Wien, Vienna, Austria
- Sejnjoen Central Hospital, Seinäjoki, Finland
- Germany (2):
  - Charité Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Leipzig, Leipzig
- Hospital Universitario Quirónsalud Madrid, Madrid, Spain
- Schulthess Klinik, Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 sites in 5 European countries. The first participant was enrolled on February 14, 2022 and the last participant had the last study visit on July 22,2022.
Pre-assignment Details: The choice of the specific BD Spinal Needle type, size, and length required for an individual participant was left to the discretion of the clinician. In this post market study, 160 participants, who were to receive a neuraxial procedures with a BD Spinal Needle as per routine clinical practice, were observed through 7-days post procedure to assess for adverse events/complications.
Groups:
- All Participants: Participants who require a BD Spinal needle as part of their routine medical care.
  Spinal needle: Insertion of a spinal needle to perform the neuraxial procedure according to the clinical practice.
Period: Overall Study
Arm/Group | All Participants
Started | 160
Enrolled Set | 160 (Participants who signed the informed consent)
Evaluable Set | 144 (Participants who underwent a neuraxial procedure, regardless of success)
Safety Set | 142 (Participants who successfully received a placement of the study device.)
Completed | 142
Not Completed | 18
Not completed — Screening Failure | 1
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — General anesthesia at the request of the surgeon | 2
Not completed — Study physician not available for the anesthesia | 3
Not completed — Anesthesia rejected by the patient on the day of surgery | 1
Not completed — Device not listed in the study was used for the procedure | 1
Not completed — Surgery not performed | 3

BASELINE CHARACTERISTICS:
Population: 160 subjects signed informed consent (Enrolled Set). 1 subject was screening failure due to "Previous spine surgery at level involved in the study procedure" and 144 subjects underwent a neuraxial procedure, regardless of success (Evaluable Set). The Evaluable set has been considered for the baseline analysis population.
Arm/Group | All Participants
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (18.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 143
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 5
  Finland | 35
  Germany | 73
  Spain | 31
Body Max Index [Mean (Standard Deviation); unit: kg/m^2] | 27.51 (4.934)
Primary diagnosis for intervention [Count of Participants; unit: Participants]
  Surgery of lower extremities | 65
  Surgery of lower abdomen | 16
  Surgery of perineum | 2
  Surgery of hips and pelvis | 9
  Obstetric | 5
  Other | 47
Reason for neuraxial procedure [Count of Participants; unit: Participants]
  Reason for neuraxial procedure:anesthesia | 144
  Reason for neuraxial procedure:analgesia | 0
  Reason for neuraxial procedure: other | 0
American Society of Anesthesiologists (ASA) physical status (PS) classification [Count of Participants; unit: Participants] — ASA I = A normal healthy patient ASA II = A patient with mild systemic disease ASA III = A patient with severe systemic disease ASA IV = A patient with severe systemic disease that is a constant threat to life
  Participants
    ASA PS Classification I | 39
    ASA PS Classification II | 82
    ASA PS Classification III | 23
Spinal needle placement details- Participant position during spinal needle procedure [Count of Participants; unit: Participants]
  Lateral position | 39
  Sitting position | 105
Spinal needle placement details - Aseptic technique [Count of Participants; unit: Participants]
  Aseptic technique = Chlorhexidine | 26
  Aseptic technique = Betadine | 6
  Aseptic technique = Other | 112
Spinal needle placement details - Local anesthesia [Count of Participants; unit: Participants]
  Local anesthesia = Lidocaine 1% | 105
  Local anesthesia = Lidocaine 2% | 5
  Local anesthesia = Other | 34
Spinal needle placement details - Lumbar interspace [Count of Participants; unit: Participants] — Lumbar interspace refers to last try with the spinal needle to achieve the spinal procedure.
  Participants
    L2-L3 | 12
    L3-L4 | 104
    L4-L5 | 27
    Other | 1
Spinal needle placement details - Number of Puncture attempts [Count of Participants; unit: Participants] — Number of puncture attempts is the number of different needles attempted to achieve the spinal procedure.
  Participants
    Number of Puncture attempts = 1 | 136
    Number of Puncture attempts = 2 | 3
    Number of Puncture attempts = 3 | 3
    Number of Puncture attempts = 4 | 2
Spinal needle placement details - Number of Interspace levels attempts [Count of Participants; unit: Participants] — The number of interspace levels attempts refers to the number of different lumbar interspace.
  Participants
    Number of Interspace levels attempts = 1 | 132
    Number of Interspace levels attempts = 2 | 10
    Number of Interspace levels attempts = 3 | 2
Spinal needle placement details - Paresthesia verbalized by participant [Count of Participants; unit: Participants]
  Paresthesia not verbalized by participant | 138
  Paresthesia verbalized by participant | 6
Spinal needle placement details - Spontaneous appearance of CSF emerging from the needle hub [Count of Participants; unit: Participants] — Number of participants with a successful needle placement in the subarachnoid space defined as the appearance of cerebrospinal fluid (CSF) from the spinal needle hub
  Participants
    Spontaneous appearance of Cerebrospinal Fluid (CSF) emerging from the needle hub | 142
    No Spontaneous appearance of Cerebrospinal Fluid (CSF) emerging from the needle hub | 2
Spinal needle placement details - BD Spinal needle type [Count of Participants; unit: Participants]
  BD Spinal Quincke needle 22Gx90mm | 5
  BD Spinal Quincke needle 27Gx90mm | 34
  BD Spinal Whitacre needle 25Gx103mm plus BD Introducer 20Gx32mm | 19
  BD Spinal Whitacre needle 25Gx90mm plus BD Introducer 20Gx32mm | 22
  BD Spinal Whitacre needle 27Gx103mm plus BD Introducer 22Gx32mm | 1
  BD Spinal Whitacre needle 27Gx90mm plus BD Introducer 22Gx32mm | 63
Spinal needle placement details - BD Syringes [Count of Participants; unit: Participants]
  BD Syringe size 5mL used | 34
  BD Syringe size 10mL used | 1
  No BD Syringe used | 109

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety: Incidence of Post-dural Puncture Headache (PDPH).
Description: Percentage of participants with a diagnosis of PDPH in the 7 days following the anesthesia procedure.
Time Frame: From insertion up to 7 days post procedure
Population: Out of 144 participants who received a neuraxial procedure, a total of 142 participants received a successful placement of the study device and were included in the safety set, used for the primary safety calculation.
Measure: Number (95% Confidence Interval); unit: % of subjects with a PDPH
Arm/Group | All Participants
Number analyzed (Participants) | 142
% of subjects with a PDPH | 2.8 [0.8 to 7.1]

2. Primary Outcome: Primary Performance: Incidence of Successful Needle Placement
Description: Successful needle placement in the subarachnoid space defined as the appearance of cerebrospinal fluid from the spinal needle hub.
Time Frame: During the insertion procedure
Population: 160 subjects signed informed consent. As 1 subject was screening failure, and for other 15 subjects a study procedure was not attempted, the study device was attempted to be placed in 144 subjects: evaluable set, used for primary performance calculation.The study device could not be placed successfully in 1 subject due to pronounced left convex scoliosis and 1 subject with successful placement was not treated via the study device.142 subjects successfully received a placement of the study device
Measure: Number (95% Confidence Interval); unit: % of successful needle placement
Arm/Group | All Participants
Number analyzed (Participants) | 144
% of successful needle placement | 98.6 [95.1 to 99.8]

3. Secondary Outcome: Secondary Safety:Incidence of Any Needle or Procedure-related Spinal/Epidural Hematoma.
Description: Incidence of device/procedure-related adverse events including the incidence of any spinal/epidural hematoma.
Time Frame: From insertion up to 7 days post procedure
Population: 160 subjects signed informed consent. As 1 subject was screening failure, and for the other 15 subjects a study procedure was not attempted, the study device was attempted to be placed in 144 subjects that constitutes the evaluable set used for secondary safety calculation.
Measure: Number (95% Confidence Interval); unit: % of subject with a spinal hematoma
Arm/Group | All Participants
Number analyzed (Participants) | 144
% of subject with a spinal hematoma | 0.0 [0.0 to 2.5]

4. Secondary Outcome: Secondary Safety: Incidence of Any Needle or Procedure-related Nerve Damage (Pain or Weakness Lower Extremities).
Description: Incidence of any device or procedure-related adverse events, including the incidence of any nerve damage (pain or weakness lower extremities).
Time Frame: From insertion up to 7 days post procedure
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: % of subject with a nerve damage
Arm/Group | All Participants
Number analyzed (Participants) | 144
% of subject with a nerve damage | 0.0 [0.0 to 2.5]

5. Secondary Outcome: Secondary Safety: Incidence of Any Needle or Procedure-related Infection (Meningitis, Spinal Abscess)
Description: Incidence of device/procedure-related adverse events including the incidence of any infection (meningitis, spinal abscess)
Time Frame: From insertion up to 7 days post procedure
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: % of subject with an infection
Arm/Group | All Participants
Number analyzed (Participants) | 144
% of subject with an infection | 0.0 [0.0 to 2.5]

6. Secondary Outcome: Secondary Safety: Incidence of Any Needle or Procedure-related Pain, Skin Redness, Irritation at or Near the Skin Puncture Site.
Description: Incidence of device/procedure-related adverse events including the incidence of any pain, skin redness, irritation at or near the skin puncture site.
Time Frame: From insertion up to 7 days post procedure
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: % subjects with pain/readness/irritation
Arm/Group | All Participants
Number analyzed (Participants) | 144
% subjects with pain/readness/irritation | 1.4 [0.2 to 4.9]

7. Secondary Outcome: Secondary Safety: Incidence of Any Needle or Procedure-related Backache.
Description: Incidence of device/procedure-related adverse events including the incidence of backache.
Time Frame: From insertion up to 7 days post procedure
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: % of subjects with backache
Arm/Group | All Participants
Number analyzed (Participants) | 144
% of subjects with backache | 0.7 [0.0 to 3.8]

8. Other Pre Specified Outcome: Spinal Needle Placement Details - Ease of Use Survey Determined by a Composite Score of BD Spinal Needle and Related Stylet Performance Based on Post-insertion Survey.
Description: After the neuraxial procedure data was recorded, the physician investigator completed a short survey to assess the performance of the BD devices used in the procedure.
  The ease-of-use survey was conducted among physician investigator to obtain information on BD spinal needle and related stylet performance.
Time Frame: After spinal needle placement
Population: 160 subjects signed informed consent. As 1 subject was screening failure, and for the other 15 subjects a study procedure was not attempted, the study device was attempted to be placed in 144 subjects that constitutes the evaluable set used for this specific measure. 143 is the overall number of subjects analyzed because 1 physician did not complete the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 143
Participants
  BD Spinal Needle insertion was easy or very easy | 135
  BD Spinal Needle withdrawal after placement was easy or very easy | 143
  PIs were agree with "stylet helped to determine the direction of spinal needle tip" | 131
  PIs were agree or strongly agree with "stylet functioned properly during spinal needle placement". | 143
  Ease of BD Stylet removal from the spinal needle after placement was easy or very easy | 142

9. Other Pre Specified Outcome: Spinal Needle Placement Details - Ease of Use Survey Determined by a Composite Score of BD Spinal Introducer Performance Based on Post-insertion Survey.
Description: After the neuraxial procedure data was recorded, the physician investigator completed a short survey to assess the performance of the BD devices used in the procedure.
  When the BD ancillary devices (e.g., spinal introducer) were used, the ease-of-use survey was conducted among physician investigator to obtain information on their performance.
Time Frame: After spinal needle placement
Population: Considering that the Spinal Introducer is an optional aid to perform the spinal procedure, 105 Introducers have been used by physicians to perform the study procedure, but only for 104 of 105 subjects for which the BD introducer has been used, the investigators completed the questionnaire and answered the respective question.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 104
Participants
  Use of the BD Introducer was easy or very easy | 104
  PIs were agree with "introducer facilitated placement of spinal needle" | 103

10. Other Pre Specified Outcome: Spinal Needle Placement Details - Ease of Use Survey Determined by a Composite Score of BD Syringe Performance Based on Post-insertion Survey.
Description: After the neuraxial procedure data was recorded, the physician investigator completed a short survey to assess the performance of the BD devices used in the procedure.
  When the BD ancillary devices (e.g., BD syringe) were used, the ease-of-use survey was conducted among physician investigator to obtain information on their performance.
Time Frame: After spinal needle placement
Population: Considering that this study is an observational study in which the physicians performed the spinal procedure according to their clinical practice and hence, they could choose any ancillary devices to achieve the study procedure, 35 BD syringes have been used by physicians to perform the study procedure, and the investigators completed the questionnaire and answered the respective question.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 35
Participants
  Reading BD Syringe graduations when preparing the dose for spinal injection was very easy | 35
  Securely connecting between the BD Syringe and the BD Spinal Needle hub was easy or very easy | 32
  Disconnecting the syringe from the spinal needle after injection was very easy | 31

ADVERSE EVENTS:
Time Frame: From the BD Spina needle insertion up to 7 days post procedure
Description: An AE is defined as any untoward medicaloccurrence, unintended disease or injury,or untoward clinical signs (includingabnormal laboratory findings) in subjects,users or other persons, whether or notrelated to the investigational medicaldevice.
  An adverse device effect is defined asany adverse event that is considered tobe related to the use of an investigationalmedical device.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/144
Serious Adverse Events (participants affected / at risk) | 0/144
Other Adverse Events (participants affected / at risk) | 17/144
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=144)
Procedural failure (General disorders) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Injection site irritation (Injury, poisoning and procedural complications) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 4 (4)
Puncture site pain (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Paresthesia (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI submits to Sponsor for review a draft 90 days prior to submission of thedraft for publication.Draft shall not divulge any confidential info.Sponsor hasthe right to:review and make comments on any proposed publication; withholdthe use of its name in connection with publication;make any results from thestudy known to its customers and governmental agencies prior topublication.The first publication of the study results shall be made inconjunction with the results from the other PIs.

DOCUMENTS (2):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT05214560/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT05214560/SAP_001.pdf